CLINICAL TRIAL: NCT03023410
Title: Using Intraoperative Sensing Technology to Evaluate Revision Total Knee Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: limited eligible population
Sponsor: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Revision TKA Study
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
Keywords: Revision TKA; Instability; Stiffness; Aseptic Loosening; Polyethylene Wear; Malrotation; Soft Tissue Imbalance
MeSH Terms: conditions — Osteoarthritis, Knee; Volvulus Of Midgut

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Partial Revision: A "partial" revision will be indicated when only the tibial liner is changed or only the tibial liner with the tibial tray or only the tibial liner with the femoral component.
  Interventions: Procedure: VERASENSE
- Total Revision: A "total" revision will be indicated when all components are completely removed and replaced (tibial tray, femoral component and tibial liner).
  Interventions: Procedure: VERASENSE

INTERVENTIONS:
Procedure: VERASENSE — Sensor-Assisted Revision TKA
  Other Names: Sensor-Assisted TKA

SUMMARY:
This study will attempt to draw relationships between the soft-tissue related complications contributing to early TKA revision and the loading and positional patterns from intraoperative tibial trial sensors. The data from the sensors may enable the surgeon to address such soft-tissue abnormalities that may otherwise be unknown during traditional total knee revision procedures. The utilization of sensors should in theory, help diagnose the potential causes attributing to soft-tissue imbalance and may lead to a decreased need for an all component revision. Furthermore, the economic implications from converting a total revision to a partial revision could have a profound effect to the patient and healthcare provider such as decreased rehabilitation regimes and opportunity for cost savings. Eligible revision patients who agree to participate will be followed for a period of 12 months following the revision procedure. Patient reported outcomes measures (PROM) such as the 2011 Knee Society Score (KSS) and the Veterans Rand 12-Item Health Survey (VR-12) will be collected at baseline (pre-operatively) and at 6 weeks, 6 months and 12 months post-procedure. All outcomes will be scored to observe changes from baseline at 12-months. Cost-analyses of sensor-assisted revision TKA will be performed to include OR costs, facility and physician fees, as well as payments to post-acute collaborators such as SNFs, rehab hospitals, PT and home care providers. A quantitative analysis of commercial payer claims / usage data (e.g., CMS Medpar data) will be used to examine costs associated with traditional revision TKA procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing revision unilateral total knee arthroplasty within the first 5-years of the index procedure
* Include Male and Female subjects
* Include subjects 18 years and older
* Patients should present with idiopathic pain and/or instability/stiffness attributed to aseptic loosening, polyethylene wear or malrotation
* Patients able to understand study intent, and agree to study participation
* Patients must be previously implanted with the following cruciate-retaining (CR) or posterior-substituting (PS) total knee systems: Stryker TRIATHLON, Zimmer-Biomet VANGUARD or NEXGEN or Smith and Nephew LEGION or JOURNEY II.

Exclusion Criteria:

* No prior revision surgery on operative side
* Ligament insufficiencies, prior surgeries such as PCL reconstructions, posterolateral reconstructions, osteotomies, tibia plateau fractures
* Culture positive aspiration indicating infection of the joint
* ASA class > III
* History of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for revision TKA and meet all inclusion and no exclusion will be offered study participation without regard to race, sex, economic status, or religious belief.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Leone, MD, Principal Investigator — Holy Cross Hospital
Locations (1):
- Holy Cross Hospital, Orthopedic Institute, Fort Lauderdale, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The investigator decided to terminate the study because the evaluable population required for the study was very limited after only one subject was recruited during the one-year recruitment period.
Period: Overall Study
Arm/Group | Partial Revision | Total Revision
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — study termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: No subject was recruited for the "Partial Revision" study arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Partial Revision | Total Revision | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: No data were collected for Sex/Gender
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cause of Early TKA Revision
Description: The objective is to evaluate and link the possible causes of early TKA revision procedures using intraoperative sensors in effort to understand why knees fail in addition to examining the economic implications to the patient and hospital.
Time Frame: 12-months
Population: 12 months follow up did not occur due to study termination
Arm/Group | Partial Revision | Total Revision
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Knee Society Score
Description: This survey is subdivided into a knee score that rates only the knee joint itself and a functional score that rates the patient's ability to walk and climb stairs. Patient expectations as well as patient satisfaction are also evaluated.
Time Frame: 12 months
Population: No outcome data was analyzed because of study termination before reaching 12 months period
Arm/Group | Partial Revision | Total Revision
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Veterans Rand 12-Item Health Survey
Description: This survey is primarily used to measure health related quality of life, to estimate disease burden and to evaluate disease-specific impact on general and selected populations. The items on the questionnaire correspond to eight principal health domains including general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue , social functioning and mental health
Time Frame: Change from Baseline at 12-months
Population: no outcome data was analyzed because of study termination before reaching 12 months period
Arm/Group | Partial Revision | Total Revision
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Date of inclusion to date of termination up to 6 months
Description: No patient was enrolled to the "partial revision" group.
Groups:
- Partial Revision: Revision of tibial liner.
- Total Revision: Revision of all components
Arm/Group | Partial Revision | Total Revision
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partial Revision (N=0) | Total Revision (N=1)
Operative site (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) — Knee pain after patient twisted operated knee
Operative site (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) — Knee pain after patient fell on the operated knee

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT03023410/Prot_SAP_000.pdf